CLINICAL TRIAL: NCT07004101
Title: Effect of Virtual Reality-based Therapy Combined With Balance Training on Biodex Balance System in Female Patients With Fibromyalgia
Brief Title: Effect of Virtual Reality Combined With Balance Training on Biodex Balance System in Female With Fibromyalgia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Dina Othman, Assisted professor, Badr University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005765
Record Dates: First submitted 2025-05-18; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Virtual Reality

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): Group ( A) will perform exercise which done by VR and biodex training
  Interventions: Other: virtual reality; Other: biodex training
- intervention (Experimental): Group (B) will perform biodex training only
  Interventions: Other: virtual reality; Other: biodex training
- conventional (Other): group (C) will perform conventional balance exercise
  Interventions: Other: conventional balance exercises

INTERVENTIONS:
Other: virtual reality — virtual reality and biodex training
  Arms: Intervention; intervention
Other: biodex training — biodex training
  Arms: Intervention; intervention
Other: conventional balance exercises — conventional balance exercises
  Arms: conventional

SUMMARY:
Is there an effect of virtual reality based therapy combined with balance training using biodex balance system on female patients with fibromyalgia .

DETAILED DESCRIPTION:
PURPOSE: To Study the Effect of virtual reality based therapy combined with balance training using biodex balance system on female patients with fibromyalgia .

BACKGROUND: Fibromyalgia (FM) is a chronic disorder defined by report of chronic widespread pain including axial pain and presence of multiple tender points on physical exam . Beyond the defining criteria.A recent survey reported balance problems as one of the top 10 most debilitating symptoms with prevalence of 45%. Balance or postural stability is a very complex task that involves the integration of multiple sensory inputs to execute appropriate neuromuscular activity needed to maintain balance .

Biodex balance system is a relatively new instrument that can be used for the assessment and management of balance dysfunction. Preliminary studies reported positive effects of balance training on Biodex balance system for the improvement of balance function.

Virtual reality based therapy (VRBT) could be effective as a non-pharmacological alternative intervention to reduce pain in women with FM. It improves dynamic balance, as it is an active therapy that requires engaging in physical activities during the sessions.VRBT requires autonomous movement of different body parts that can increase muscle tone and the perception of pain-free movement favoring the elimination of restrictions to movement included in the cerebral body scheme due to continued pain.

ELIGIBILITY:
Inclusion Criteria:

* Women patients from age 35 to 50 years old
* All patients describe a history of pain spreading in all quadrants of the body for at least three months and pain is caused by digital pressure in at least 11 out of 18 allogenic points, called tender points

Exclusion Criteria:

* Old neglected fracture
* Malignant diseases
* Neurological diseases.
* Uncontrolled diabetes

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
BIODEX BALANCE ASSESMENT | pre and post treatment 4 weeks
  BIODEX used to asses balance

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt